CLINICAL TRIAL: NCT06424522
Title: Low Anterior Resection Syndrome: Retrograde Enema Program vs Medical Management
Brief Title: A Bowel Management Program (Retrograde Rectal Enema) for the Treatment of Low Anterior Resection Syndrome in Rectal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Alessandra, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-22312; NCI-2024-03173 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Low Anterior Resection Syndrome; Rectal Carcinoma
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms | interventions — Dietary Fiber; Enema; Loperamide; Physical Therapy Modalities; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (RRE, medical management) (Experimental): Patients undergo a bowel management program comprising a medical management pathway (fiber, loperamide hydrochloride, pelvic floor physical therapy) in combination with RRE treatment for 1 year. Patients use the RRE system to self administer an individualized enema regimen via the rectum. Patients may undergo abdominal film x-rays throughout the trial.
  Interventions: Dietary Supplement: Dietary Fiber; Procedure: Enema Administration; Drug: Loperamide Hydrochloride; Procedure: Physical Therapy; Other: Questionnaire Administration; Procedure: X-Ray Imaging
- Group II (medical management) (Active Comparator): Patients receive medical management comprising fiber, loperamide hydrochloride, and pelvic floor therapy for 1 year. If medical management fails, patients may then be referred for surgery with sacral nerve stimulator placement.
  Interventions: Dietary Supplement: Dietary Fiber; Drug: Loperamide Hydrochloride; Procedure: Physical Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Dietary Fiber — Receive dietary fiber
  Other Names: Fiber
Procedure: Enema Administration — Undergo RRE
  Other Names: Enema; Enema Injection
  Arms: Group I (RRE, medical management)
Drug: Loperamide Hydrochloride — Receive loperamide hydrochloride
  Other Names: Imodium; Imodium A-D
Procedure: Physical Therapy — Undergo pelvic floor physical therapy
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure
Other: Questionnaire Administration — Ancillary studies
Procedure: X-Ray Imaging — Undergo abdominal film x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; Static X-Ray; X-Ray
  Arms: Group I (RRE, medical management)

SUMMARY:
This clinical trial studies if a bowel management program with a retrograde rectal enema (RRE) for the treatment of low anterior resection syndrome (LARS) in rectal cancer patients is better than medical management alone. Rectal cancer treatment can include a procedure where part of the rectum with cancer is removed and the remaining part of the rectum is reconnected to the colon, this is called a low anterior resection of the rectum. LARS is a common condition that can develop after undergoing a low anterior resection of the rectum. LARS consists of any change in how the body performs defecation, the discharge of feces from the body, after undergoing a resection procedure. Patients with LARS may experience fecal urgency, incontinence, increased frequency, constipation, feelings of incomplete bowel movement, or bowel emptying difficulties. Patients may experience individual symptoms of LARS or a combination of them. A bowel management program assists patient's with identifying a specific bowel management regimen that works best for managing symptoms of LARS. A RRE consists of inserting a catheter through the anus into the rectum. The RRE is designed to assist fecal emptying. Medical management of LARS can include the use of fiber, loperamide hydrochloride, or pelvic floor physical therapy. Fiber may help relieve constipation, feelings of incomplete bowel movement, or bowel emptying difficulties. Loperamide hydrocholoride may help lessen fecal urgency, incontinence, or increased frequency. Pelvic floor physical therapy may help restore strength in the rectum possibly helping to improve symptoms of LARS. Participating in a bowel management program with a RRE may be more effective in treating LARS than medical management alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare two approved pathways for treatment of low anterior resection syndrome (LARS) - a retrograde enema program versus a medical management pathway.

SECONDARY OBJECTIVE:

I. The determination of feasibility to complete this treatment pathway.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo a bowel management program comprising a medical management pathway (fiber, loperamide hydrochloride, pelvic floor physical therapy) in combination with RRE treatment for 1 year. Patients use the RRE system to self administer an individualized enema regimen via the rectum. Patients may undergo abdominal film x-rays throughout the trial.

GROUP II: Patients receive medical management comprising fiber, loperamide hydrochloride, and pelvic floor therapy for 1 year. If medical management fails, patients may then be referred for surgery with sacral nerve stimulator placement.

Upon completion of study intervention all patients are followed up at 1 month, 3 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Moderate to Severe LARS diagnosis
* Patients with history of rectal cancer that was treated with proctectomy
* Has undergone standard medical management without improvement of symptoms for 3-6 months

Exclusion Criteria:

* Patients presenting with significant stricture that need a definitive surgical management strategy; patients with minor or clinically negligible strictures can still be candidates. Patients who are able to pass the catheter and the balloon per rectum may be candidates after a digital rectal exam at their initial visit
* Patients with any chemo or radiation therapy in the last 6 months
* Patients who currently have colorectal cancer
* Patients with recurrent colorectal cancer
* Patients who have undergone a colorectal surgical procedure within the last three months
* Patients with progressive neurological disease
* Patients with active or recurrent sacral infection
* Patients < 18 years old
* Active sacral nerve simulator
* Pregnant or planning to become pregnant during the treatment portion of the study
* Altered mental status or mental disability that would alter ability to self-administer enema
* Any reason the research team believes the subject is not an appropriate candidate for this study (i.e., transportation issues, history of no-show appointments, lack of reliable communications, vulnerable population(s), etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Fecal incontinence | Up to 1 year from start of treatment
  Will be measured using a validated scoring tool for LARS (Memorial Sloan Kettering Cancer Center Bowel Function Instrument Questionnaire [MSKCC BFI]). Effect size (Cohen's d > 0.80) will be computed to ensure the effect of findings. P < 0.05 is considered significant. Statistical analysis will be conducted using linear or nonlinear mixed modelling as found appropriate by the statistician.
Effectiveness assessed using LARS validated scoring tool | Up to 1 year from start of treatment
  Will be assessed using LARS validated scoring tool. Effect size (Cohen's d > 0.80) will be computed to ensure the effect of findings. P < 0.05 is considered significant. Statistical analysis will be conducted using linear or nonlinear mixed modelling as found appropriate by the statistician.

SECONDARY OUTCOMES:
Feasibility measured by Patient Satisfaction Survey | At 1 year from start of treatment
  Will be assessed by administering a patient satisfaction survey post treatment. Effect size (Cohen's d > 0.80) will be computed to ensure the effect of findings. P < 0.05 is considered significant. Statistical analysis will be conducted using linear or nonlinear mixed modelling as found appropriate by the statistician.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra C Gasior, DO, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu